CLINICAL TRIAL: NCT03871348
Title: A Phase 1 First-in-Human Dose Escalation and Expansion Study for the Evaluation of Safety, Pharmacokinetics, Pharmacodynamics and Anti-tumor Activity of SAR441000 Administered Intratumorally as Monotherapy and in Combination With Cemiplimab in Patients With Advanced Solid Tumors
Brief Title: A First-in-Human Dose Escalation and Expansion Study to Evaluate Intratumoral Administration of SAR441000 as Monotherapy and in Combination With Cemiplimab in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated the study for non-safety reasons
Sponsor: Sanofi (Industry)
Collaborators: BioNTech RNA Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED15297; U1111-1205-1176 (Registry Identifier: ICTRP); 2017-004766-94 (EudraCT Number)
Record Dates: First submitted 2019-01-24; First posted 2019-03-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- SAR441000 Dose Escalation Phase (Experimental): SAR441000 will be administered as intratumoral injection as monotherapy in patients with solid tumors over a 28-day cycle
  Interventions: Drug: SAR441000
- SAR441000 + cemiplimab - Dose Escalation Phase (Experimental): SAR441000 will be administered as intratumoral injection in patients with solid tumors in combination with cemiplimab over a 21-day cycle
  Interventions: Drug: SAR441000; Drug: Cemiplimab REGN2810
- SAR441000 + cemiplimab Expansion Melanoma, anti-PD-1 failure (Experimental): SAR441000 will be administered intratumorally at the determined recommended dose in combination with cemiplimab to patients with advanced melanoma who have failed anti-PD-1/PD-L1 therapy. Treatment is administered over a 21-day cycle
  Interventions: Drug: SAR441000; Drug: Cemiplimab REGN2810
- SAR441000 + cemiplimab Expansion Melanoma, anti-PD-1 naive (Experimental): SAR441000 will be administered intratumorally at the determined recommended dose in combination with cemiplimab to patients with advanced anti-PD-1/PD-L1 naïve melanoma over a 21-day cycle
  Interventions: Drug: SAR441000; Drug: Cemiplimab REGN2810
- SAR441000 + cemiplimab Expansion CSCC, anti-PD-1 naive (Experimental): SAR441000 will be administered intratumorally at the determined recommended dose in combination with cemiplimab to patients with advanced anti-PD-1/PD-L1 naïve Cutaneous Squamous Cell Carcinoma (CSCC) over a 21-day cycle
  Interventions: Drug: SAR441000; Drug: Cemiplimab REGN2810
- SAR441000 + cemiplimab Expansion HNSCC, anti-PD-1 naive (Experimental): SAR441000 will be administered intratumorally at the determined recommended dose in combination with cemiplimab to patients with advanced anti-PD-1/PD-L1 naïve Head and Neck Squamous Cell Cancer (HNSCC) over a 21-day cycle
  Interventions: Drug: SAR441000; Drug: Cemiplimab REGN2810

INTERVENTIONS:
Drug: SAR441000 — Pharmaceutical form: concentrate for solution for injection
  Route of administration: intratumoral
Drug: Cemiplimab REGN2810 — Pharmaceutical form: solution for injection
  Route of administration: intravenous
  Arms: SAR441000 + cemiplimab - Dose Escalation Phase; SAR441000 + cemiplimab Expansion CSCC, anti-PD-1 naive; SAR441000 + cemiplimab Expansion HNSCC, anti-PD-1 naive; SAR441000 + cemiplimab Expansion Melanoma, anti-PD-1 failure; SAR441000 + cemiplimab Expansion Melanoma, anti-PD-1 naive

SUMMARY:
Primary Objectives:

* Dose Escalation: To determine maximum tolerated dose (MTD) or maximum administered dose (MAD) and overall safety and tolerability profile of SAR441000 when administered intratumorally as monotherapy and in combination with cemiplimab in patients who have no alternative standard treatment options.
* Dose Expansion (Combination): To determine the objective response rate of SAR441000 administered intratumorally in combination with cemiplimab in patients with melanoma, cutaneous squamous cell carcinoma or head and neck squamous cell carcinoma.

Secondary Objectives:

* To characterize the pharmacokinetic (PK) profile of SAR441000 administered as monotherapy and in combination with cemiplimab.
* To assess the immunogenicity of SAR441000.
* To characterize the safety of SAR441000 when administered intratumorally in combination with cemiplimab.
* To determine the disease control rate (DCR), duration of response (DoR) and progression free survival (PFS) of SAR441000.
* To determine the recommended dose of SAR441000 for the expansion phase.

DETAILED DESCRIPTION:
The expected duration of treatment for patients who benefit from study intervention may vary, based on progression date. Median expected duration of study per patient is estimated as 9 months in monotherapy and 12 months in combination therapy.

The maximum treatment duration for non-progressive patients is up to 2 years.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age
* Advanced solid tumors including lymphomas for which no standard alternative therapy is available (escalation phase).
* Advanced melanoma (Stage IIIB-C or Stage IV, anti-PD-1/PD-L1 treated or not) or anti-PD-1/PD-L1 not treated advanced Head and Neck Squamous Cell Cancer or anti-PD-1/PD-L1 not treated Advanced Cutaneous Squamous Cell Cancer where no other alternative treatment option exists (expansion phases).
* Minimum 3 lesions enrollment.
* Injectable disease (i.e., suitable for direct intratumoral injection based on the dose level volume of each cohort and cumulative lesion size; according to the investigator's judgement).
* A lesion amenable for additional tumor biopsy.
* Patients with measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Life expectancy more than 3 months.
* Willingness to provide mandatory tumor biopsy.
* Male and female patients who agree to use effective contraceptive methods.
* Signed informed consent.

Exclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance score >1.
* Significant and uncontrolled concomitant illness that would adversely affect the patient's participation in the study.
* Any prior organ transplantation.
* History within the last 5 years of an invasive malignancy other than the one treated in this study, with the exception of resected basal or squamous-cell skin cancer or carcinoma, in situ of cervix or other local tumors considered cured by local treatment.
* History of unresolved viral hepatitis; systemic immune suppression including acquired immunodeficiency syndrome (AIDS) related illnesses or human immunodeficiency virus (HIV) disease requiring antiretroviral treatment.
* Prior splenectomy.
* New and progressive brain lesions.
* Poor bone marrow reserve resulting in low blood cell count.
* Poor liver and kidney functions, abnormal coagulation tests.
* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments.
* Maintenance therapy with prednisolone >7.5 mg/day orally or equivalent during the study.
* Non-resolution of any prior treatment related toxicity to Grade <2, except alopecia, vitiligo, fatigue and hypothyroidism controlled with replacement therapies.
* Moderate to severe immune related adverse event to prior immune-modulating agents within 90 days prior to the first study treatment.
* Central nervous system lymphoma.
* Prior allogeneic hematopoietic stem cell transplantation (HSCT) for patients with lymphoma.
* Autologous HSCT less than 90 days prior to initiation of study intervention.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
For dose escalation: Incidence of Dose Limiting Toxicities (DLTs) (Monotherapy) | Cycle 1; Cycle = 28 days for monotherapy
  Incidence of DLTs at Cycle 1 (SAR441000 monotherapy), assessed as the occurrence of AE, satisfying protocol defined DLT criteria, using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 whether related or not to the study treatment in the absence of clear evidence to the contrary, and if not related to a disease progression
For dose escalation: Incidence of Dose Limiting Toxicities (DLTs) (Combination therapy) | Cycle 1 Day 1 to Cycle 2 Day 8; Cycle = 21 days for combination therapy; overall assessment = 28 days
  Incidence of DLTs during period from Cycle 1 Day 1 to Cycle 2 Day 8 (SAR441000 + cemiplimab combination therapy), assessed as the occurrence of AE, satisfying protocol defined DLT criteria, using NCI-CTCAE version 5.0 whether related or not to the study treatment in the absence of clear evidence to the contrary, and if not related to a disease progression
For dose escalation: Maximum tolerated dose (MTD) of SAR441000 (Monotherapy) | End of Dose Escalation phase (ie, End of Cycle 1 for last patient); Cycle = 28 days for monotherapy
  MTD of SAR441000 as monotherapy, determined during Cycle 1 of dose escalation phase
For dose escalation: Maximum tolerated dose (MTD) of SAR441000 (Combination therapy) | End of Dose Escalation Phase (ie, End of Cycle 1 Day 1 to Cycle 2 Day 8 for last patient); Cycle = 21 days for combination; overall assesment = 28 days
  MTD of SAR441000, in combination with cemiplimab, determined during period from Cycle 1 Day 1 to Cycle 2 Day 8 in dose escalation phase
Adverse Events | Up to end of treatment (Estimated median duration=12 months)
  Incidence of Treatment Emergent Adverse Events (TEAE) during dose escalation phase
For Expansion: Objective Response Rate (ORR) | Estimated median duration = 12 months
  Assessment of overall response rate using standard imaging and RECIST 1.1 criteria

SECONDARY OUTCOMES:
Assessment of Pharmacokinetic (PK) parameter for SAR441000 (Cmax) (Monotherapy) | Cycle 1 Week 1 and Cycle 3 Week 1 (in all patients); Cycle duration is 28 days for monotherapy
  Maximum plasma concentration (Cmax) of SAR4410000 as monotherapy observed over the dosing interval
Assessment of Pharmacokinetic (PK) parameter for SAR441000 (Cmax) (Combination therapy) | Cycle 1 Week 1 and Cycle 3 Week 1 (in all patients); Cycle duration is 21 days for combination therapy
  Maximum plasma concentration (Cmax) of SAR4410000 in combination with cemiplimab observed over the dosing interval
Assessment of PK parameter for SAR441000 (AUC) (Monotherapy) | Cycle 1 Week 1 and Cycle 3 Week 1 (in all patients); Cycle duration is 28 days for monotherapy
  Area under the plasma concentration versus time curve (AUC) of SAR441000 as monotherapy over the dosing interval
Assessment of PK parameter for SAR441000 (AUC) (Combination therapy) | Cycle 1 Week 1 and Cycle 3 Week 1 (in all patients); Cycle duration is 21 days for combination therapy
  Area under the plasma concentration versus time curve (AUC) of SAR441000 in combination with cemiplimab over the dosing interval
Assessment of PK parameter (Ctrough) for SAR441000 | Baseline to End of Treatment (Estimated median duration of 12 months)
  Trough Plasma Concentration (Ctrough) of SAR441000 as monotherapy and in combination with cemiplimab. It is defined as plasma concentration observed just before treatment administration during repeated dosing
Assessment of PK parameter for cemiplimab (Cmax) | Cycle 1; Cycle duration is 21 days
  Maximum plasma concentration of cemiplimab in combination with SAR441000, observed over the dosing interval
Assessment of PK parameter of cemiplimab (AUC) | Cycle 1; Cycle duration is 21 days
  Area under the plasma concentration versus time curve of cemiplimab in combination with SAR441000 over the dosing interval
Assessment of PK parameter for cemiplimab (Ctrough) | Baseline to End of Treatment (Estimated median duration of 12 months)
  Trough plasma concentration of cemiplimab in combination with SAR441000, observed just before treatment administration during repeated dosing
Immunogenicity of SAR441000 and cemiplimab | Baseline to End of Study (Estimated median duration of 12 months)
  Incidence of anti-drug antibody (ADA) positive patients for immunogenicity
DCR | Baseline to End of Study (Estimated median duration of 12 months)
  Disease Control Rate (DCR) with SAR441000 in combination with cemiplimab. DCR is sum of Complete Response + Partial Response + Stable Disease
DoR | Baseline to End of Study (Estimated median duration of 12 months)
  Duration of Response (DoR) with SAR441000 in combination with cemiplimab. DoR is time from initial response to the first documented tumor progression
Progression Free Survival (PFS) | Baseline to End of Study (Estimated median duration of 12 months)
  Time from first drug administration to the first documented tumor progression or death from any cause, whichever comes first
Incidence of Treatment Emergent Adverse Events (TEAE) during dose expansion phase | Baseline to End of Treatment (Estimated median duration of 12 months)
  Incidence of Adverse Events (AE)/ Serious AE (SAE) / Laboratory abnormalities considered to be adverse events
Recommended dose of SAR441000 for expansion phase (Combination therapy) | End of Dose Escalation Phase (ie, End of Cycle 1 Day 1 to Cycle 2 Day 8 for last patient); Cycle = 21 days for combination; overall assesment = 28 days
  SAR441000 dose for administration in combination with cemiplimab selected for expansion phase based on MTD/MAD by the Bayesian model, the overall safety, activity and PK/PDy data
For Dose Expansion: Objective Response Rate (ORR) | Estimated median duration of 12 months
  Assessment of overall response rate using standard imaging by RECIST 1.1 and iRECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (19):
- United States (3):
  - Dana-Farber Cancer Institute- Site Number : 8400003, Boston, Massachusetts
  - Cleveland Clinic - Cleveland- Site Number : 8400007, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center- Site Number : 8400002, Houston, Texas
- Belgium (3):
  - Investigational Site Number : 0560001, Brussels
  - Investigational Site Number : 0560003, Ghent
  - Investigational Site Number : 0560002, Leuven
- France (3):
  - Investigational Site Number : 2500004, Marseille
  - Investigational Site Number : 2500002, Paris
  - Investigational Site Number : 2500001, Villejuif
- Germany (5):
  - Investigational Site Number : 2760005, Hamburg
  - Investigational Site Number : 2760004, Heidelberg
  - Investigational Site Number : 2760001, Mainz
  - Investigational Site Number : 2760003, Mannheim
  - Investigational Site Number : 2760006, Tübingen
- Netherlands (2):
  - Investigational Site Number : 5280002, Nijmegen
  - Investigational Site Number : 5280001, Rotterdam
- Spain (3):
  - Investigational Site Number : 7240004, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240001, Pamplona, Navarre
  - Investigational Site Number : 7240002, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Bechter O, Loquai C, Champiat S, Baurain JF, Grob JJ, Utikal J, Rottey S, Berrocal A, Hassel JC, Arance A, Sanmamed MF, Boers-Sonderen M, Gastman B, Gebhardt C, Delafontaine B, Sahin U, Tureci O, Brueck P, Abbadessa G, Marpadga R, Lee H, Yang Y, Buday B, Di Genova G, Wang H, Xia B, Lee JS, Lebbe C. A Phase I, First-in-Human, Dose-Escalation, Expansion Trial of Cytokine-Encoding Synthetic mRNA Mixture Alone or with Cemiplimab in Advanced Solid Tumors. Clin Cancer Res. 2025 Jun 13;31(12):2358-2369. doi: 10.1158/1078-0432.CCR-24-1983. PMID 40152791
- See also: TED15297 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25356&tenant=MT_SNY_9011